CLINICAL TRIAL: NCT04817774
Title: Multicentre Open-Label Single Ascending Dose Dose-Ranging Phase I/IIa Study to Evaluate Safety and Tolerability of an Autologous Antigen-Specific Chimeric Antigen Receptor TRegulatory Cell Therapy in Living Donor Renal Transplant Recipients
Brief Title: Safety & Tolerability Study of Chimeric Antigen Receptor T-Reg Cell Therapy in Living Donor Renal Transplant Recipients
Acronym: STEADFAST
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sangamo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: TX200 KT02; 2019-001730-34 (EudraCT Number); 2024-512579-11-00 (EU CTIS Number)
Record Dates: First submitted 2021-03-09; First posted 2021-03-26 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Kidney Transplant Rejection; End Stage Renal Disease
Keywords: Regulatory T cells; Genetically modified cells; Chimeric Antigen Receptor; Living donor; Autologous
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Subjects undergo kidney transplant as per planned standard of care and are administered study drug post transplantation.
  Interventions: Biological: TX200-TR101
- Control group and Transplant donors (No Intervention): Control group: Subjects undergo kidney transplant as per planned standard of care with no study drug administered.
  Transplant donors: Transplant donors for each subject in the treatment and control groups.

INTERVENTIONS:
Biological: TX200-TR101 — TX200-TR101 is an autologous gene therapy medicinal product composed of Treg cells (CD4+/CD45RA+/CD25+/CD127low/neg) that have been ex vivo expanded and transduced with a lentiviral vector encoding for a CAR to recognize HLA-A*02. Treatment will be given via an IV infusion at a pre-defined timepoint several weeks after transplant. Four, single ascending dose cohorts of TX200-TR101 are planned and an additional expansion cohort.
  Other Names: CAR-Tregs
  Arms: Treatment group

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of TX200-TR101 and its effects on the donated kidney in living donor kidney transplant recipients. TX200-TR101 is a product made from a kidney transplant recipient's own immune cells, which are genetically modified and designed to help the transplant recipient's body accept their donated kidney and prevent their immune system from rejecting it.

DETAILED DESCRIPTION:
This is a multicentre, first-in-human, open-label, single ascending dose, dose-ranging study of autologous, chimeric antigen receptor T regulatory cells (CAR-Treg) in HLA-A2 mismatched living donor kidney transplant recipients, with a control cohort of mismatched kidney transplant recipients of similar immunological risk.The aim is for the CAR-Tregs to recognise the HLA-A2 molecule present on the donated kidney and subsequently induce and maintain immunological tolerance to the organ.

The study requires three different types of participants - transplant recipients who will receive the study treatment TX200-TR101; control participants, who are transplant recipients who will not receive the study treatment; and transplant donors, who will donate their kidney to the transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Male or female aged 18 - 70 years.
* Diagnosis of End Stage Renal Disease and waiting for a new kidney from an identified live donor.
* Subjects who will be single organ recipients (kidney).
* Able and willing to use contraception.

Exclusion Criteria:

* HLA identical to the donor.
* Subjects with prior organ transplant.
* Known hypersensitivity to study medication ingredients, protocol defined immunosuppressive medications, or a significant allergic reaction to any drug.
* Positive serology for human immunodeficiency virus (HIV) or syphilis, active or occult hepatitis B virus (HBV), active hepatitis C virus (HCV) infection, or other clinically active local or systemic infection.
* Subjects who are Epstein-Barr Virus (EBV) seronegative.
* Positive flow cytometric crossmatch using donor lymphocytes and recipient serum.
* Subjects with panel-reactive antibody (PRA) >20% within 6 months prior to enrolment.
* Subjects with current or recent donor-specific antibodies.
* Use of any experimental medicinal product within 3 months.
* Current use of systemic immunosuppressive agents
* Significant unstable or poorly controlled acute or chronic diseases (except ESRD), limited life expectancy, clinically relevant central nervous system pathology, history of drug/alcohol abuse or psychiatric disorder or other condition that is not compatible with adequate study follow-up, history of malignancy in the past 5 years and any other reason that, in the opinion of the Site Investigator or Medical Monitor, would render the subject unsuitable for participation in the study.
* Subjects with abnormal laboratory values in the following parameters:
* Haemoglobin
* Platelets
* White blood cells
* Aspartate transaminase (AST) and or alanine transaminase (ALT)
* Total bilirubin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women of childbearing potential: negative pregnancy test
Enrollment: 26 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2025-10-29 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 28 days post infusion
  Safety and tolerability of TX200-TR101 infusion evaluated by incidence and grade of treatment-emergent adverse events (TEAEs), including serious adverse events (SAEs) according to CTCAE V5.0.

SECONDARY OUTCOMES:
Acute graft related outcomes | Day of infusion through to Week 84
  Incidence of biopsy confirmed acute rejection according to the Banff classification criteria
Long-term safety | Day of infusion through to Week 84
  Number of transplant recipient subjects with TEAEs, including SAEs, as assessed by CTCAE v5.0
Immunosuppression | Day of infusion through to Week 84
  Ability to reduce immunosuppression as measured by the proportion of subjects receiving tacrolimus monotherapy at Week 84
Graft localization | Day of infusion through to Week 84
  Graft localization of TX200-TR101 cells as measured by the presence of CD4+ CAR+ cells in the renal transplant biopsy
Chronic graft related outcomes | Day of infusion through to Week 84
  Chronic graft dysfunction as measured by estimated glomerular filtration rate
Chronic graft related outcomes | Day of infusion through to Week 84
  Incidence of chronic graft rejection according to the Banff criteria for chronic rejection

CONTACTS AND LOCATIONS:
Locations (5):
- University Hospitals Leuven, Leuven, Belgium
- Netherlands (3):
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Centre, Leiden
  - Erasmus MC, University Medical Center, Rotterdam
- Oxford University Hospitals NHS Foundation Trust,, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No